CLINICAL TRIAL: NCT02278835
Title: To Analyze the Effectiveness of Respiratory Physiotherapy Techniques in the Post Operative Mitral Valve
Brief Title: The Effectiveness of Respiratory Physiotherapy in Mitral Valve Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Maria Ignez Zanetti Feltrim, Drª Maria Ignez Zanetti Feltrim, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAPPesq 0011/09
Record Dates: First submitted 2014-10-02; First posted 2014-10-30 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Mitral Valve Disease
Keywords: Cardiac valve
MeSH Terms: interventions — Breathing Exercises; Intermittent Positive-Pressure Breathing; Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- level1 (Other): Patients classified in level 1 were randomized in the breathing exercises group or incentive spirometry group
  Interventions: Other: breathing exercises; Device: incentive spirometry
- level2 (Other): Patients classified in level 2 were randomized in the Intermittent Positive Pressure Breathing group or Continuous Positive Airway Pressure group
  Interventions: Device: Intermittent positive pressure breathing; Device: Continuous positive airway pressure

INTERVENTIONS:
Other: breathing exercises — 3 sets of 10 repetitions of deep breathing exercises
  Other Names: EXE
  Arms: level1
Device: incentive spirometry — 3 sets of 10 repetitions of deep breathing exercises with incentive spirometry
  Other Names: IS (Coach®)
  Arms: level1
Device: Intermittent positive pressure breathing — 20 minutes breathing with intermittent positive pressure
  Other Names: IPPB (BIRD Mark 7™)
  Arms: level2
Device: Continuous positive airway pressure — 20 minutes breathing with continuous positive airway pressure
  Other Names: CPAP (Sullivan®)
  Arms: level2

SUMMARY:
This trial was conducted to evaluate the effectiveness of the chest physiotherapy techniques to prevent pulmonary collapse based in an score applied in the patients submitted of the mitral valve surgery, after their ICU discharge.

Patients were allocated in groups according their pulmonary function (FVC: forced vital capacity), the respiratory muscle performance (MIP: maximal inspiratory pressure; MEP: maximal expiratory pressure), the oxygenation level (SpO2), the pulmonary auscultation; respiratory frequency (f); the ability to expectorate and the functional independence.

The group I was allocated those patients which presented decrease of up to 50% of forced vital capacity (FVC) of preoperative period, SpO2>92%, minimal pulmonary auscultation alterations; frequency (f) between 15 and 25 ipm; able to expectorate without assistance; independence to sit; respiratory. In these patients were randomized for two interventions: a) Deep breathing exercises: diaphragmatic exercises; inspiratory sighs; maximal inspiration exercises. Each kind of exercises was repeated 10 times; b) volume-targeted incentive spirometer: used Coach® three sets of 10 repetitions.

Patients allocated in the group II presented FVC> 30% <49% of preoperative period, ≥ 88% SpO2 <92%, necessity of oxygen therapy, abnormal pulmonary auscultation, f> 25 <31ipm; dependence to expectorate and to sit.. They were assisted by: a) Intermittent Positive Pressure Breathing (IPPB) with PEEP - through ventilator (Bird Mark 7™) with exhalation valve spring load set at 10 cmH2O. b) CPAP - 10 cmH2O associated with oxygen support to obtain SpO2≥ 95% with electronic device (Sullivan®) Each session consisted of 20 minutes, twice daily, one in the morning and another in the afternoon.

All of the patients were conducted in effort to mobilize upper and lower limbs. On the first day, the patients walked at least 50 meters, by increasing the distance to at least 150 meters on the fourth day. Outcome measures were recorded at day 5 of the interventions.

DETAILED DESCRIPTION:
The study were conducted with individuals of both gender, aged between 18 and 60 years, candidates for mitral valve surgery, up to a maximum 2nd valve replacement. Patients unable to perform the functional tests were excluded and patients with signs of neurological disorders; hemodynamic instability, respiratory disorders and mechanically ventilated for more than 48 hours .

ELIGIBILITY:
Inclusion Criteria:

* Patients for mitral valve surgery, up to a maximum 2nd valve replacement

Exclusion Criteria:

* Patients unable to perform the functional tests
* Patients with signs of neurological disorders; hemodynamic instability, respiratory disorders and mechanically ventilated for more than 48 hours

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2009-03; Primary Completion 2014-01 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
incidence of atelectasis | Patients were followed for five days

SECONDARY OUTCOMES:
pulmonary function | Patients were followed for five days
  Forced vital capacity in liters and percentual (FVC; %FVC )
pulmonary function | Patients were followed for five days
  Forced expiratory volume in first second in liters and percentual (FEV1; %FEV1)
pulmonary function | Patients were followed for five days
  Ratio of forced expiratory volume in first second and forced vital capacity (FEV1/FVC)

OTHER OUTCOMES:
Respiratory Muscle Strength | Patients were followed for five days
  Maximum inspiratory pressure (MIP)
Respiratory Muscle Strength | Patients were followed for five days
  Maximum expiratory pressure (MEP)

REFERENCES:
- [Background] Matte P, Jacquet L, Van Dyck M, Goenen M. Effects of conventional physiotherapy, continuous positive airway pressure and non-invasive ventilatory support with bilevel positive airway pressure after coronary artery bypass grafting. Acta Anaesthesiol Scand. 2000 Jan;44(1):75-81. doi: 10.1034/j.1399-6576.2000.440114.x. PMID 10669276
- [Result] Pasquina P, Tramer MR, Walder B. Prophylactic respiratory physiotherapy after cardiac surgery: systematic review. BMJ. 2003 Dec 13;327(7428):1379. doi: 10.1136/bmj.327.7428.1379. PMID 14670881